CLINICAL TRIAL: NCT00326365
Title: A Multicenter, Randomized, Double Blind, Placebo Controlled Trial to Investigate the Efficacy and Safety of the Homeopathic Remedy Kalium Bichromicum (Potassium Dichromate) to Decrease Viscosity and Amount of Sputum as Well as Time to Extubation, in Intubated Mechanically Ventilated ICU Patients.
Brief Title: Effect of Homeopathic Remedy Kalium Bichromicum on Viscosity and Amount of Sputum Mechanically Ventilated ICU Patients.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KAL.ICU.2006
Record Dates: First submitted 2006-05-15; First posted 2006-05-16 (Estimated); Last update posted 2007-10-31 (Estimated); Status verified 2006-05

CONDITIONS: Mechanically Ventilated ICU Patients
Keywords: mechanical ventilation; secretions; viscosity; homeopathy; kalium bichromate; extubation

INTERVENTIONS:
Drug: Kali bichromicum 10-60 (C30)

SUMMARY:
The purpose of this study is to determine whether the homeopathic remedy Kali Bichromium is effective in reducing the amount of tracheal secretions in patients intubated with a conventional endotracheal tube and receiving controlled mechanical ventilation in the ICU setting.

DETAILED DESCRIPTION:
Profuse and tenacious tracheal secretions are a significant factor impeding the weaning process in mechanically ventilated patients in the intensive care unit (ICU). In homeopathy, high dilutions of plant extracts, minerals, and other biological substances are used as remedies for the treatment of illness, which is based on the "Law of Similars" (the higher the dilution, the stronger the effect). Kali Bichromicum (potassium dichromate) is a drug that is commonly used in homeopathy, mostly for conditions involving profuse, stringy, tenacious mucous and tracheal secretions. A recent randomized, double-blind, placebo-controlled study found a statistically significant effect of this remedy on improving the amount of tracheal secretion, timing to extubation and discharge from the ICU among critically ill patients, with no side effects observed.

The proposed study will compare the efficacy of Kali bichromicum 10-60 (C30) versus placebo in reducing the amount of tracheal secretions in patients intubated with a conventional endotracheal tube and receiving controlled mechanical ventilation in the ICU setting. Both the quantity and viscoelasticity (measured by rheometry) of the secretions will be studied, as well as sputum neutrophil count (using direct microscopy). Time to extubation and the need for re-intubation will also be evaluated. 56 patients over the age of 18 years treated with mechanical ventilation for at least 3 days will be recruited from the ICU departments of 4 medical centers in Israel. The preparations will be administered in the form of small pellet-like globules, which will be placed on the mucosa of the mouth, to the side of the endotracheal tube. Patients will be randomly allocated to either verum (n=28) or placebo (n=28) treatment, with the remedies administered twice daily with an interval of 12 hours, for a period of up to 14 days or until the patient is extubated. Any adverse event will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. any endotracheally intubated ICU patient on mechanical ventilation support for at least 3 days prior to study enrollment.
2. profuse tenacious, stringy tracheal secretions

Exclusion Criteria:

* Unstable septic patients
* Concomitant disease of the larynx and trachea obstructing the airway or inhibiting the extubation process.
* Patients with Tracheostomy
* Concomitant active heart disease.
* Need for catecholamines.
* Pregnancy.
* Patient with underlying neuromuscular disorder or any other condition preventing patient cooperation with voluntary coughing and expectoration of secretions.
* Patients with underlying conditions requiring continuous therapy with bronchorrheic medications (i.e. myasthenia gravis)
* Failure of the patient or legal guardian to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2006-06

PRIMARY OUTCOMES:
To compare efficacy of Kali bichromicum (C30) in reducing tracheal secretions in mechanically ventilated patients

SECONDARY OUTCOMES:
To compare the proportion of patients with grade 3 tracheal secretions;number of suctionings;reduction of tracheal secretions;effects on the mucus viscoelasticity and sputum neutrophil count; shortening time to extubation and need for re-intubation.
effect in shortening the time to discharge from the ICU. To evaluate the safety of of Kali bichromicum 10-60 (C30) as compared with placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Menachem Oberbaum, M.D., Principal Investigator — Shaare Zedek Medical Center, Jerusalem, Israel
Locations (1):
- Intensive Care Unit, Shaare Zedek Medical Center, Jerusalem, Israel

REFERENCES:
- [Background] Frass M, Dielacher C, Linkesch M, Endler C, Muchitsch I, Schuster E, Kaye A. Influence of potassium dichromate on tracheal secretions in critically ill patients. Chest. 2005 Mar;127(3):936-41. doi: 10.1378/chest.127.3.936. PMID 15764779